CLINICAL TRIAL: NCT06245083
Title: Evaluating Pyrroloquinoline Quinone (PQQ) for Improving Obese Pregnancy Outcomes (EPyQ)
Brief Title: Evaluating Pyrroloquinoline Quinone (PQQ) for Improving Obese Pregnancy Outcomes
Acronym: EPyQ
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Investigator did not return submission for final IRB approval. Study was withdrawn by IRB.
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 16843
Record Dates: First submitted 2024-01-10; First posted 2024-02-07 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Maternal Obesity
MeSH Terms: conditions — Pregnancy in Obesity | interventions — PQQ Cofactor; Soybean Oil

STUDY DESIGN:
Intervention Model Description: Participants are randomized to receive either pyrroloquinoline quinone (PQQ) or placebo
Who Masked: Participant, Investigator
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- PQQ supplement (Active Comparator): Pyrroloquinoline quinone (PQQ) 20 mg/day
  Interventions: Drug: Pyrroloquinoline quinone (PQQ)
- Placebo (Placebo Comparator): Placebo supplement with soybean oil 20 mg/day
  Interventions: Drug: Placebo with soybean oil

INTERVENTIONS:
Drug: Pyrroloquinoline quinone (PQQ) — Oral supplement taken daily
  Arms: PQQ supplement
Drug: Placebo with soybean oil — Oral supplement taken daily
  Arms: Placebo

SUMMARY:
Maternal obesity (MO) affects 1 in 5 women and is strongly linked to increased birth weight, childhood/adolescent obesity, life-long metabolic and inflammatory disorders, and childhood neuropsychiatric disorders. There remains a critical unmet need for developing a safe and effective non-pharmacological approach for attenuating metabolic inflammation and ameliorating the adverse effects of MO on offspring health that originate in utero and extend into the lactational period. Pyrroloquinoline quinone (PQQ) is a diet-derived natural food supplement with anti-inflammatory properties that, in humans and mice, improves metabolism and exerts potent immunoregulatory effects. Researchers' central hypothesis is that PQQ administration during MO pregnancy 1) improves maternal metabolic and inflammatory indices, 2) improves utero-placental blood flow and ameliorates placental maladaptation (oxidative stress, hypoxia, inflammation and fatty acid transporter expression) and 3) reduces neonatal adiposity.

DETAILED DESCRIPTION:
Women with a body mass index (BMI) greater than 30 will be recruited during their first trimester clinic visit up to 16 weeks of gestation. In addition to the blood draw and anthropometric measurements normally carried out at the first pre-natal visit, researchers will provide consented study subjects with pyrroloquinoline quinone (PQQ) or placebo in capsules at a dose of 20 milligrams per day. There will be 15 women per group. At ~30 days after initiating the study (4-week routine follow-up visit) blood samples will be obtained. At ~24-28 weeks gestation, during the 2nd trimester visit, study subjects will undergo the standard 1-hour oral glucose screen, routine prenatal complete blood count (CBC) evaluation, study maternal blood sampling, and anthropometric measurements. During the delivery inpatient admission, researchers will again collect maternal blood as well as placental tissue, and umbilical cord blood (plasma, aperipheral blood mononuclear cells) after delivery. Placental tissue (samples from four separate cotyledons) will be collected for protein (homogenate and plasma membrane isolation), ribonucleic acid (RNA), quantitative polymerase chain reaction (qPCR), and histology (fixed in 4% paraformaldehyde). The neonate will undergo PeaPod evaluation prior to discharge, and within 72 hours after birth. PQQ supplementation will continue for 30 days post-partum at which time maternal blood and breastmilk samples will be collected, as well as a follow up infant Peapod evaluation and maternal dual x-ray absorptiometry (DEXA) scan.

ELIGIBILITY:
Inclusion Criteria:

* Adult women
* Body mass index >30 kg/m2
* Currently pregnant with gestational age up to 16 wks

Exclusion Criteria:

* Women with pregestational diabetes (type 1 or type 2)
* Smokers
* Women with other risk factors for placental insufficiency or preterm delivery
* Advanced maternal age (age ≥40 yrs)
* Pre-existing chronic hypertension
* Renal disease
* Thrombophilias
* Substance use
* Human immunodeficiency virus (HIV)
* Hepatitis C
* Autoimmune disorders

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only pregnant adult women will be recruited for this study.
Enrollment: 0 (Actual)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Leptin | 1 month postpartum
  Measured at multiple time points from maternal blood samples
Adiponectin | 1 month postpartum
  Measured at multiple time points from maternal blood samples
Triglycerides (TGs) | 1 month postpartum
  Measured at multiple time points from maternal blood samples
High-density lipoprotein cholesterol (HDL-C) | 1 month postpartum
  Measured at multiple time points from maternal blood samples
Low-density lipoprotein cholesterol (LDL-C) | 1 month postpartum
  Measured at multiple time points from maternal blood samples
Very-low-density lipoprotein cholesterol (VLDL-C) | 1 month postpartum
  Measured at multiple time points from maternal blood samples
C-reactive protein (CRP) | 1 month postpartum
  Measured at multiple time points from maternal blood samples
Soluble CD163 (sCD163) | 1 month postpartum
  Measured at multiple time points from maternal blood samples
Lipopolysaccharides (LPS) | 1 month postpartum
  Measured at multiple time points from maternal blood samples
Glucose | 24-28 weeks
  Measured from routine gestational diabetes screening
Infant fat mass | 1-3 days postpartum
  Measured using air-displacement plethysmography (PEAPODTM)
Infant fat-free mass | 1-3 days postpartum
  Measured using air-displacement plethysmography (PEAPODTM)
Infant weight | 1-3 days postpartum
  Measured using scale
Infant body length | 1-3 days postpartum
  Measured using measuring tape or board
Infant limb length | 1-3 days postpartum
  Measured using measuring tape or board
Infant head circumference | 1-3 days postpartum
  Measured using measuring tape
Infant abdominal circumference | 1-3 days postpartum
  Measured using measuring tape
Infant chest circumference | 1-3 days postpartum
  Measured using measuring tape
Infant mid-thigh circumference | 1-3 days postpartum
  Measured using measuring tape
Infant mid-arm circumference | 1-3 days postpartum
  Measured using measuring tape

CONTACTS AND LOCATIONS:
Overall Officials: Marty Maxted, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No